CLINICAL TRIAL: NCT04715243
Title: Comparison of High Flow Nasal Cannula (HFNC), Face-mask Non-Invasive Ventilation (NIV) & Helmet NIV in COVID-19 ARDS Patients
Acronym: NIV COVID19
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 1. Futility
  2. Lack of recruitment in the centers due to lack of cases meeting the study criterial despite period of extension.
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Abdulhakeem Al-Hashim, Senior Consultant, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SQU-EC/206/2020
Record Dates: First submitted 2021-01-09; First posted 2021-01-20 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Acute Respiratory Distress Syndrome Caused by COVID-19

STUDY DESIGN:
Intervention Model Description: Multi-centre randomized trial of confirmed COVID-19 cases presenting to the emergency department, the ward, high dependency or intensive care unit (ICU) with ARDS requiring non-invasive mechanical ventilation. They will be assigned to one of the three arms; high flow nasal cannula (HFNC), Face-mask NIV or Helmet NIV.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control (Other): Face-mask NIV is the standard of care
  Interventions: Device: Face-mask NIV
- intervention 1 (Active Comparator): High flow nasal cannula
  Interventions: Device: High flow nasal cannula (HFNC)
- Intervention 2 (Active Comparator): Helmet NIV
  Interventions: Device: Helmet NIV

INTERVENTIONS:
Device: High flow nasal cannula (HFNC) — High flow nasal cannula as a form of non-invasive oxygen delivery
  Arms: intervention 1
Device: Helmet NIV — NIV interface
  Arms: Intervention 2
Device: Face-mask NIV — NIV interface
  Arms: control

SUMMARY:
Objective: To determine whether NIV delivered through helmet interface reduces intubation rate among patients with COVID-19 ARDS compared to face-mask NIV and HFNC.

Design, setting & participants: Two-center randomized clinical trial of 360 patients with mild to moderate ARDS and confirmed COVID-19 requiring non-invasive ventilation between August 2020 to January 2021. The patients with respiratory rate (RR) more than 30/min or oxygen saturation (SpO2) less than 90% or PaO2/FiO2 ratio less than 300 despite standard oxygen therapy by face mask (<15 L/min) who present to Royal hospital or Sultan Qaboos University Hospital (SQUH) emergency department, medical wards or intensive care unit (ICU).

Intervention: Patients will be randomly assigned (block randomization) to either face-mask NIV, HFNC or Helmet NIV. The helmet is a transparent hood that covers the entire head of the patient and has a rubber collar neck seal.

Main outcome and measures: The primary outcome is the rate of endotracheal intubation at 28-days. Secondary outcomes include hospital mortality at 28 and 90 days, NIV free days, invasive ventilator free days and hospital length of stay.

Expected results: We assume the failure rate of Helmet NIV to be 30%, failure rate of HFNC to be 40% and failure rate of face-mask NIV to be 50%. A sample size of 360 patients (120/group) will achieve a power of 0.90 at a significance level of 0.05. To account for 10% dropout rate, the total sample required is 396 subjects(132/group).

DETAILED DESCRIPTION:
Inclusion criteria:

* > 18 years of age
* confirmed COVID-19
* Within 48 hours of presentation in the emergency department, high dependency area or intensive care unit (ICU)
* ARDS according to Berlin definition (P/F < 300) or O2 saturation < 90% or RR > 30/min) in room air
* Standard oxygen therapy at flow rate < 15L/min x 60 minutes

Exclusion criteria:

* More than 48 hours of admission to the emergency room, high dependency or intensive care unit
* On non-invasive ventilation or HFNC for more than 4 hours before enrollement
* Impending cardiopulmonary arrest
* Need for immediate endotracheal intubation
* Hemodynamic instability or life-threatening arrhythmias
* GCS < 8
* Active intracranial pathology or high ICP
* Inability to cooperate or protect the airway
* Pregnancy
* Tracheostomy
* DNR or refusing intubation
* Known type 2 respiratory failure
* On chronic home oxygen therapy

Enrolment:

Multi-centre randomized trial of confirmed COVID-19 cases presenting to the emergency department, the ward, high dependency or intensive care unit (ICU) with ARDS requiring non-invasive mechanical ventilation. It is an open label randomized clinical trial. We will perform permuted block randomization of 9 and perform concealment.

Consent:

A written consent must be taken from the patient or the decision maker prior to enrollment.

Each of the three arms have pre-specified treatment protocol in the form of algorithm.

For the helmet NIV group, for type 1 respiratory failure (hypoxemia & normal pCO2), CPAP will be started at 10 cmH2O & FiO2 0.6. Re-assessment will be done every 15-30 minutes and CPAP and FiO2 will be increased accordinly (CPAP to 15 & FiO2 of 1.0 maximum) If patients develops hypercapnia, the mode will be changed to BiPAP: IPAP 12-25 cmH2O (max 20) EPAP 8-15 cmH2O.

In the face-mask NIV group, CPAP will be started at 5 cmH2O & FiO2 0.6. Re-assess will be performed every15-30 minutes. Thereafter CPAP & FiO2 will be adjusted accordingly (maximum CPAP 12 & FiO2: 1.0) If the patient develops high pCO2 :BiPAP: IPAP 8-20 cmH2O (max 20) EPAP 4-12 cmH2O.

In the high flow nasal cannula group, HFNC will be started at at 20-30 L/min Adjust FiO2 to keep SpO2 > 92%. Thereafter, it will be titrated to flow to max 60 L/min & FiO2 100%

For all the three groups, these are the following targets:

Target:

SPO2 ≥ 92 % RR ≤ 30/min ROX index > 2.85 at 2 hours and > 3.85 at 12 hours (HFNC group)

If the above targets are not achieved, the ICU team will assess them for possible endotracheal intubation. In case the patient doesn't tolerate any of the two NIV interfaces, they will be allowed to cross over to the other with intention to treat analysis. For the high flow oxygen group, a trial of non-invasive ventilation will be allowed at the physician discretion before endotracheal intubation with intention to treat analysis.

Statistical Analysis:

We tested the null hypothesis that there is no difference between the Helmet-NIV, HFNC and face-mask-NIV intubation rate and the alternative hypothesis that Helmet NIV and HFNC is superior to face-mask-NIV. We assumed the failure rate of Helmet NIV to be 30% and the failure rate of HFNC to be 40% and failure rate of face-mask NIV is 50%. The group subject counts are allocated 1:1:1. The effect size is 0.12. A sample of 360 subjects, (120/group) achieves a power of 0.90 at a significance level of 0.05. To account for 10% dropout rate, the total sample required is 396 subjects(132/group).

Baseline characteristics will be reported by mean and standard deviation for the continuous variables and numbers and proportions for categorical variables. Intention to treat analysis to analysis will be used for the results for the primary efficacy point of reduction in the rate of the intubation between the three groups. Fisher's exact test will be used between-group differences in the rate of intubation. The face-mask-NIV is considered as a control group as it is the standard treatment and will calculate t the relative risk and absolute risk difference for the primary end points. The log-rank test will compare the time from enrollment to ET intubation for the three groups using Kaplan-Meier curves plot. Similar analysis will be performed for the 28-day mortality for as the secondary end points. All P values reported for on primary and secondary end points are based on two-sided tests of 0.05. The SAS statistical software is used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* confirmed COVID-19
* Within 48 hours of presentation in the emergency department, high dependency area or intensive care unit (ICU)
* ARDS according to Berlin definition (P/F < 300) or O2 saturation < 90% or RR > 30/min) in room air
* Standard oxygen therapy at flow rate < 15L/min x 60 minutes

Exclusion Criteria:

* More than 48 hours of admission to the emergency department, high dependency or intensive care unit
* More than 4 hours on NIV or HFNC before enrolment
* Impending cardiopulmonary arrest
* Need for immediate endotracheal intubation
* Hemodynamic instability or life-threatening arrhythmias
* GCS < 8
* Active intracranial pathology or high ICP
* Inability to cooperate or protect the airway
* Pregnancy
* Tracheostomy
* DNR or refusing intubation
* Known type 2 respiratory failure
* On chronic home oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Rate of endotracheal intubation | within the study period with an average of one month.
  The patient will be randomly assigned to one of the treatment arms. Then the patient will be followed up for one month for the primary outcome which is endotracheal intubation.

SECONDARY OUTCOMES:
Hospital mortality | 90 days from the hospital mortality.
  Number of patients who survived compared to who died in each intervention
Hospital length of stay | Throughout the study completion. An average of 90 days.
  total number of days patients remain in the hospital as inpatient in each intervention
Ventilator free days | Throughout the study completion. An average of 90 days.
  number of days patients remain off intervention (invasive or non-invasive)

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan Qaboos University Hospital, Muscat, Oman

IPD SHARING:
Plan to Share IPD: Yes
Publish in a journal
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after July 2021

REFERENCES:
- [Derived] Al Hashim AH, Al Reesi A, Al Lawati NM, Burad J, Al Khabori M, Chandwani J, Al Lawati R, Al Masroori Y, Al Balushi AA, Al Masroori S, Al Siyabi K, Al Lawati F, Ahmed FYN, Al Busaidy M, Al Huraizi A, Al Jufaili M, Al Zaabi J, Varghese JT, Al Harthi R, Sebastian KP, Al Abri FH, Al Aghbari J, Al Mubaihsi S, Al Lawati A, Al Busaidi M, Foti G. Comparison of Noninvasive Mechanical Ventilation With High-Flow Nasal Cannula, Face-Mask, and Helmet in Hypoxemic Respiratory Failure in Patients With COVID-19: A Randomized Controlled Trial. Crit Care Med. 2023 Nov 1;51(11):1515-1526. doi: 10.1097/CCM.0000000000005963. Epub 2023 Jun 13. PMID 37310174